CLINICAL TRIAL: NCT04134650
Title: Effect of Low Dose Combination of Linagliptin and Metformin to Improve Pancreatic Beta Cell Function, Insulin Resistance and Cardiovascular Function in Patients With Prediabetes and Overweight/Obesity: Randomizer Clinical Trial
Brief Title: Effect of Low Dose Combination of Linagliptin + Metformin to Prevent Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Rodolfo Guardado Mendoza, Principal Investigator, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CI/HRAEB/2018/0018
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Prediabetic State; Insulin Resistance
Keywords: Prediabetes
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Linagliptin; Metformin

STUDY DESIGN:
Intervention Model Description: 1:1 ratio allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Medications in both groups will be supplied in identical envelopes and by a person not involved in the study. Persons involved in the follow-up and outcomes measurements will be masked to the patient´s treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linagliptin + Metformin plus lifestyle (Experimental): Patients are randomized to receive for 12 months Linagliptin 2.5mg + metformin 1700mg every 24 hours. The start of the dose in this group will be gradual so that at the month of treatment the patient can be with the full doses. Together with this, patients will receive a lifestyle modification program seeking to reduce 5-7% of body weigh and increase physical activity to 90-150min/week.
  Interventions: Combination Product: Linagliptin + metformin
- Metformin plus lifestyle (Active Comparator): Patients are randomized to receive for 12 months Metformin 1700mg every 24 hours. The start of the dose in this group will be gradual so that at the month of treatment the patient can be with the full doses. Together with this, patients will receive a lifestyle modification program seeking to reduce 5-7% of body weigh and increase physical activity to 90-150min/week.
  Interventions: Drug: Metformin

INTERVENTIONS:
Combination Product: Linagliptin + metformin — Linagliptin-Metformin 2.5/1700mg daily plus a lifestyle modification program based on nutritional assesment, physical activity prescription and general counseling
  Other Names: low doses of Linagliptin + metformin
  Arms: Linagliptin + Metformin plus lifestyle
Drug: Metformin — Metformin 1700mg daily plus a lifestyle modification program based on nutritional assesment, physical activity prescription and general counseling
  Arms: Metformin plus lifestyle

SUMMARY:
Type 2 diabetes is a chronic disease that has reached global epidemic proportions due to the growing number of patients in all countries; It has become the disease that causes more chronic and acute complications to patients, unfortunately, when the diagnosis of type 2 diabetes is made patients are identified at very advanced stages of the disease.

For all the above, the best strategies will be those that are aimed at early stages of the disease, and the investigators are convinced that the use the combination of drugs with additive pathophysiological effect plus cardiovascular protection in early stages, will have better results, lasting and with greater results impact on the natural history of the disease that throws measures that may have an applicability in clinical practice, in order to contribute to the control of this pathology. Therefore, the combination of medications with different mechanisms of action, in low doses, could be a useful strategy not only to prevent type 2 diabetes, but also to prevent macro and microvascular complications early. The goal of this clinical trial is to evaluate the effect of low doses of linagliptin + metformin vs metformin alone on physiopathological parameters, such as glucose metabolism, insulin resistance, insulin secretion and pancreatic beta cell function in patients with impaired fasting glucose plus impaired glucose tolerance, during 12 months.

DETAILED DESCRIPTION:
The main goal of this clinical trial is to compare the effect of two different treatments during 12 months:

1. Lifestyle modification program + metformin 1700mg every 24 hours.
2. Lifestyle modification program + linagliptin (2.5mg) and metformin (1700mg) every 24 hours.

on the following parameters, after 12 months of treatment:

1. Glucose metabolism, evaluated by the oral glucose tolerance
2. Insulin resistance, evaluated by the oral glucose tolerance in 100% of the patients
3. Insulin secretion, evaluated by the oral glucose tolerance in 100% of the patients
4. Pancreatic beta cell function, evaluated by the oral glucose tolerance in 100% of the patients
5. Cardiovascular function, evaluated by ejection fraction measurement, diastolic and systolic preloads measured by standard echocardiography.

All the patients will have a basal evaluation with an oral glucose tolerance test, lipid profile, body composition. After the basal evaluation, if the patients result with prediabetes (FASTING IMPAIRED GLUCOSE/IMPAIRED GLUCOSE TOLERANCE) and have at least 2 risk factors, they will be invited to the intervention phase where they will be randomized to one of the two treatment groups.

Patients will have a follow-up visit every month to review the adherence to the lifestyle modification program and to the medication. After 6 months, patients will repeat the same evaluation performed as the basal evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prediabetes, defined for the existence of one or both of the following conditions: 1) impaired fasting glucose (Fasting glucose between 100 and 125 mg/dL), 2) impaired glucose tolerance (Glucose between 140 and 199 mg/dL at the 2 hours of the Oral Glucose Tolerance test (OGTT)
* Patients who accept to participate in the study and sign the informed consent letter.

Exclusion Criteria:

* Patients with diagnosed Type 2 Diabetes Mellitus previously or detected during the OGTT
* Patients in actual treatment or during the last 3 months with metformin, pioglitazone or another antidiabetic drug, including insulin.
* Serum creatinine > 1.6 mg/dL
* Hypertriglyceridemia very high (>500 mg/dL)
* Pregnant women
* Altered arterial hypertension (Systolic > 180 mmHg or Diastolic >105 mmHg)
* Excessive alcohol intake, acute or chronic
* Medications or medical conditions that affect glucose homeostasis (thiazides, beta blockers, glucocorticoids for systemic use, weight-reducing drugs or anorexigenics, Cushing's syndrome, Thyrotoxicosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from basal fasting and 2 hours glucose levels during the oral glucose tolerance test at 12 months | 12 months
  Fasting and post-2 hours glucose values (mg/dl) during the oral glucose tolerance test

SECONDARY OUTCOMES:
Change from basal pancreatic beta cell function at 12 months | 12 months
  Evaluated with the Disposition index (DI), obtained from measurements of glucose and insulin during the oral glucose tolerance test. A higher value in the DI meas a better pancreatic beta cell function. There are not minimum and maximum levels
Change from basal insulin sensitivity at 12 months | 12 months
  Insulin sensitivity evaluated with the Matsuda Index, obtained with the insulina and glucose measurements during the oral glucose tolerance test. Matsuda index is reported in arbitrary units, and a higher value means a better insulin sensitivity. There are not minimum and maximum levels

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Guardado-Mendoza, MDPhD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanauato, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz LO, Bennett PH, Ravussin E, Kidd JR, Kidd KK, Esparza J, Valencia ME. Effects of traditional and western environments on prevalence of type 2 diabetes in Pima Indians in Mexico and the U.S. Diabetes Care. 2006 Aug;29(8):1866-71. doi: 10.2337/dc06-0138. PMID 16873794
- [Background] DeFronzo RA, Bonadonna RC, Ferrannini E. Pathogenesis of NIDDM. A balanced overview. Diabetes Care. 1992 Mar;15(3):318-68. doi: 10.2337/diacare.15.3.318. PMID 1532777
- [Background] Faerch K, Borch-Johnsen K, Holst JJ, Vaag A. Pathophysiology and aetiology of impaired fasting glycaemia and impaired glucose tolerance: does it matter for prevention and treatment of type 2 diabetes? Diabetologia. 2009 Sep;52(9):1714-23. doi: 10.1007/s00125-009-1443-3. Epub 2009 Jul 10. PMID 19590846
- [Result] Hsu SM, Raine L, Fanger H. Use of avidin-biotin-peroxidase complex (ABC) in immunoperoxidase techniques: a comparison between ABC and unlabeled antibody (PAP) procedures. J Histochem Cytochem. 1981 Apr;29(4):577-80. doi: 10.1177/29.4.6166661.
- [Result] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Result] Haffner SM, Lehto S, Ronnemaa T, Pyorala K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in nondiabetic subjects with and without prior myocardial infarction. N Engl J Med. 1998 Jul 23;339(4):229-34. doi: 10.1056/NEJM199807233390404. PMID 9673301

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04134650/Prot_SAP_000.pdf